CLINICAL TRIAL: NCT00198614
Title: A Comparison of the Effectiveness of Carvedilol Versus Metoprolol for Atrial Fibrillation Appearing After Off-Pump Coronary Bypass Surgery in the Carvedilol or Metoprolol Post-Revascularization Atrial Fibrillation Controlled Trial (COMPACT)
Brief Title: Carvedilol Versus Metoprolol for the Prevention of Atrial Fibrillation After Off-Pump Coronary Bypass Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ministry of Health, Labour and Welfare, Japan (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 16C-9
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2007-03-01 (Estimated); Status verified 2007-02

CONDITIONS: Coronary Disease; Atrial Fibrillation
Keywords: Adrenergic beta-Antagonists; Carvedilol; Metoprolol; Coronary Artery Bypass; Atrial Fibrillation
MeSH Terms: conditions — Coronary Disease; Atrial Fibrillation

INTERVENTIONS:
Drug: Carvedilol versus Metoprolol

SUMMARY:
Postoperative new-onset atrial fibrillation (AF) is the most common complication stemming from coronary artery bypass graft surgery, and is associated with increased early and late mortality risk. Standard guidelines recommend β blockers for the prevention of AF; however, no prospective study has compared the relative efficacy of β-blocking agents. We hypothesize that carvedilol, a non-selective adrenergic blocker with both anti-inflammatory and antioxidant properties, is more effective than metoprolol, a conventional β1-selective antagonist, in suppressing new-onset AF following off-pump coronary bypass surgery. We have designed the Carvedilol or Metoprolol Post-Revascularization Atrial Fibrillation Controlled Trial (COMPACT) to test our hypothesis in a multi-center, open-label, and randomized controlled trial.

DETAILED DESCRIPTION:
Occurring in 20% to 50% of patients, postoperative new-onset atrial fibrillation (AF) is the most common complication of coronary artery bypass graft (CABG) surgery. Reports have indicated that the occurrence of postoperative AF is associated with a prolonged stay in the hospital, readmission to the intensive care unit, stroke, and, consequently, increased overall costs. Moreover, recent results from both retrospective and prospective observational studies suggest that its associated early and late mortality risk is high. During the past decade, off-pump coronary bypass (OPCAB) surgery has gained widespread acceptance as an alternative to conventional on-pump CABG surgery, as avoiding cardiopulmonary bypass and myocardial ischemia-reperfusion is thought to significantly reduce postoperative systemic complications. Nevertheless, recent studies have revealed that OPCAB surgery does not reduce the incidence of postoperative AF, possibly because the consistent inflammatory differences between on-pump CABG and OPCAB surgery are present only at the beginning of the postoperative course, or partially because general surgical trauma may play a greater role. It has thus been anticipated that, as with on-pump CABG surgery, OPCAB surgery has high AF-related mortality and morbidity risks, and the prevention of new-onset AF following OPCAB surgery should significantly reduce the risk of these outcomes. To date, most reviews reflect a growing consensus in favor of the prophylactic administration of β blockers. In addition, the American College of Cardiology/American Heart Association guidelines for CABG surgery recommend β blockers for the prevention of AF. To the best of our knowledge, however, no prospective study has evaluated the merits of a specific β-blocking agent or concluded that each of these agents is equally efficacious.

Carvedilol, a non-selective beta adrenergic blocking agent approved for use in heart failure cases, has a number of ancillary activities including anti-inflammatory and antioxidant properties. Although the exact pathophysiology of new-onset AF following OPCAB surgery has not yet been elucidated, recent reports suggest that markers of inflammation and oxidative injury are elevated in patients with non-surgical AF. In addition, clinical studies indicate that, unlike the β1-selective agent metoprolol, carvedilol has incremental benefits for AF management in heart failure patients. The anti-inflammatory and antioxidant properties of carvedilol have generated interest in its use as a prophylaxis for postoperative AF.

These considerations led to the organization of COMPACT, a multi-center, randomized controlled trial of 650 patients designed to test the hypothesis that carvedilol is more effective than metoprolol, a conventional β1-selective antagonist, in suppressing new-onset AF following OPCAB surgery.

ELIGIBILITY:
Inclusion criteria:

Adult male or female patients are required to meet the following criteria:

1. Aged 20 to 89 years
2. Underwent isolated off-pump coronary artery bypass graft surgery
3. Written informed consent

Exclusion criteria:

Patients with the following conditions will be excluded from the study:

1. Pre- and intraoperative use of mechanical circulatory support devices, except an intra-aortic balloon pump
2. Concomitant operations, such as aneurysmectomy or carotid endarterectomy
3. Surgical approaches other than a median full sternotomy
4. Acute myocardial infarction ≦3 days before enrollment in the trial
5. Contraindication against treatment with β blockers
6. Presence of preoperative chronic AF or flutter
7. History of paroxysmal AF
8. Presence of antidysrhythmic medication other than β blockers, calcium channel blockers, or digitalis
9. A resting heart rate of less than 50 beats/min in the absence of medical therapy known to slow the sinus rate
10. Endocrine disorders, such as pheochromocytoma, active hyperthyroidism, and untreated hypothyroidism
11. Pregnant women and females with childbearing potential unless utilizing adequate contraception
12. Preoperative need for a temporary or permanent pacemaker
13. Non-interpretable electrocardiogram for P wave assessment
14. Undergoing treatment for asthma or other chronic obstructive pulmonary disease
15. Second- or third-degree atrioventricular block
16. Sick sinus syndrome
17. Uncontrolled heart failure
18. Unstable insulin-dependent diabetes mellitus
19. Steroid therapy requirement
20. History of autoimmune diseases
21. Active infectious diseases, including myocarditis or pericarditis
22. Any other serious disease that could potentially complicate the management and follow-up protocols

Ages: 20 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 650
Dates: Start 2005-01

PRIMARY OUTCOMES:
The primary endpoint is the incidence of new-onset AF during the first seven days after surgery; AF is defined as an episode of atrial fibrillation or flutter lasting for >30 seconds as detected on the continuous cardiac monitor.

SECONDARY OUTCOMES:
the incidence, duration, and recurrence of new-onset AF after surgery and before hospital discharge
the frequency of external or internal electrical cardioversion after surgery and before hospital discharge
the incidence of AF rhythm at hospital discharge
premature discontinuation of assigned drug administration
in-hospital mortality for any cause after surgery
in-hospital morbidity after surgery
resource use after surgery until hospital discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Masakazu Kuro, M.D., Ph.D., Principal Investigator — Department of Anesthesiology, National Cardiovascular Center
Locations (1):
- National Cardiovascular Center, Suita, Osaka, Japan